CLINICAL TRIAL: NCT02080559
Title: A Randomised, Descriptive, Open Label, Study Exploring the Relationship Between Gene Expression Signatures With Reactogenicity and Immunogenicity Following Vaccination With Serogroup B Meningococcal Vaccine (4CMenB)
Brief Title: Investigating the Immune Response to 4CMenB in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Public Health England (Other Government); Imperial College London (Other); Novartis Vaccines (Industry); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OVG2012/05 EUCLIDS
Record Dates: First submitted 2014-02-17; First posted 2014-03-06 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-02

CONDITIONS: Meningitis
MeSH Terms: conditions — Meningitis | interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4CMenB - Test group (Experimental): Administered at 2, 4 and 12 months of age
  Interventions: Biological: 4CMenB
- 4CMenB - control group (Active Comparator): Given at 5, 7 and 13 months of age
  Interventions: Biological: 4CMenB

INTERVENTIONS:
Biological: 4CMenB — 0.5ml IM
  Other Names: Bexsero

SUMMARY:
This randomised, open-label, single-centre, descriptive study aims to investigate gene expression (i.e what genes are 'switched on' and 'off') following vaccination with 4CMenB and to relate this to vaccine reactions and to immune response.

160 healthy Caucasian infants aged 8-12 weeks (at time of first visit) who have not yet received their routine infant immunisations will be recruited. Participation in the study will be limited to to Caucasian infants (defined as having two Caucasian parents). This is so that baseline variability in gene expression data which is to some degree affected by ethnicity is reduced.

Participants will be randomised to either a 'test' group or 'control' group depending on what 4CMenB schedule they receive, with 80 infants in each.

All participants will receive the usual paediatric immunisations according to the UK national immunisation schedule. In addition, participants in the test groups will receive 4CMenB at 2, 4 and at 12 months while those in the control groups will receive the same vaccine at 5, 7 and 13 months. Blood samples will be taken from each infant at specified time points before and after vaccination to address the objectives of the study.

In addition, oro-pharyneal swabs will be obtained around different vaccination timepoints to investigate the effect of 4CMenB vaccination on the oro-pharyngeal Neisseria microbiome.

DETAILED DESCRIPTION:
The incidence of meningococcal disease is 0.2-14 per 100,000 in industrialized countries. In England and Wales, during the period 2005-2010, there were 900-1300 cases annually. Disease is commonest in infants, young children and adolescents and case fatality is high at 8-10%.

Until recently there were no licensed vaccines against serogroup B meningococcal disease, although vaccines against epidemic strains of MenB have been used in several countries.

Unfortunately, 4CMenB is associated with significant reactogenicity. This is presumably related to the presence of various bacterial surface components present in the outer membrane vessicles (OMVs), including lipopolysacchride (LPS), which are capable of activating the innate immune response. The host pathways responsible for reactogenicity to OMV vaccines, and indeed to other vaccines, are not yet established, and the relationship between reactogenicity and immunogenicity is not clear.

This study will provide information about pathways and mechanisms of immunity and may identify gene expression signals which can be used in future vaccine design and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of two Caucasian parents (self-defined by parent) born between 37 and 42 weeks of gestation aged 8-12 weeks at time of first visit
* Parent or legal guardian willing and able to comply with the requirements of the protocol and have internet access for the duration of the study.
* Parent/legal guardian who have given informed consent for their child's participation in the study

Exclusion Criteria:

* Non-Caucasian infants
* Children of parents who are on the delegation log for this study
* Parent/ legal guardian under the age of 18
* History of invasive meningococcal B disease
* Previous vaccination with meningococcal serogroup B vaccine
* History of being a household contact with a case of confirmed bacterial meningitis
* Prior administration of any vaccine or planned administration of any vaccine not specified in the study protocol, with the exception of Hepatitis B vaccine and Influenza vaccines (which can be given 14 days before or after study vaccines), or BCG (which can be administered 28 days before or after study vaccines)
* Prior or planned receipt of any other investigational vaccine or drug
* Confirmed or suspected immunodeficiency
* A family history of congenital or hereditary immunodeficiency, or maternal HIV
* Receipt of more than 1 week of immunosuppressants or immune modifying drugs (e.g. oral prednisolone >0.5ml/kg/day or intravenous glucocorticoid steroid).
* History of allergy to any component of the vaccine
* Major congenital defects or serious chronic illness
* History of any neurologic disorders or seizures
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period
* Any other condition which, in the opinion of the investigator, may interfere with the ability to fulfil study requirements (this may include plans to move house and language comprehension).
* No internet access for the duration of the study.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Gene expression in whole blood at 4hr, 24hr, 3d and 7d time points following 4CMenB and routine infant vaccination given at 2, 4 and 12 months. | 13 months
  This is a descriptive study that aims to identify what genes are 'turned on' or 'turned off' following vaccination with 4CMenB and routine vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, PhD, Principal Investigator — Oxford Vaccine Group, University of Oxford
Locations (1):
- Oxford Vaccine Group, Centre for Clininal Vaccinology & Tropical Medicine, Oxford, United Kingdom

REFERENCES:
- [Derived] O'Connor D, Pinto MV, Sheerin D, Tomic A, Drury RE, Channon-Wells S, Galal U, Dold C, Robinson H, Kerridge S, Plested E, Hughes H, Stockdale L, Sadarangani M, Snape MD, Rollier CS, Levin M, Pollard AJ. Gene expression profiling reveals insights into infant immunological and febrile responses to group B meningococcal vaccine. Mol Syst Biol. 2020 Nov;16(11):e9888. doi: 10.15252/msb.20209888. PMID 33210468